CLINICAL TRIAL: NCT03786419
Title: Phase II Study to Evaluate the Efficacy and Safety of Atezolizumab in Subjects With Unresectable or Advanced Malignant Pleural Mesothelioma Who Experienced Progression on Platinum-Based Chemotherapy
Brief Title: A Study of Atezolizumab in Unresectable or Advaced Malignant Pleural Mesothelioma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Publication of study results of ICI use in MPM as first line therapy
Sponsor: Health Pharma Professional Research (Other)
Responsible Party: Principal Investigator, Jorge Arturo Alatorre Alexander, Principal Investigator, Health Pharma Professional Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JCJ-768883
Record Dates: First submitted 2018-12-18; First posted 2018-12-26 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Malignant Pleural Mesothelioma, Advanced; Malignant Pleural Mesothelioma, Unresectable
Keywords: Malignant Pleural Mesothelioma; Atezolizumab; Thoracic neoplasms; Antibodies, monoclonal; Antineoplasic, agents
MeSH Terms: conditions — Mesothelioma, Malignant; Thoracic Neoplasms | interventions — atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab (Experimental): Participants with unresectable or advanced malignant pleural mesothelioma who have progressed after platinum-based chemotherapy will receive atezolizumab 1200 mg every 21 days, until Investigator-assessed loss of clinical benefit, unacceptable toxicity, investigator or participant's decision to withdraw from therapy, or death (whichever occurs first).
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Participants will be given 1200 mg of Atezolizumab as single agent by IV infusion every 21 days. First infusion will be over 60 min. Subsequent Atezolizumab cycles may be administered for 30 minutes, if there were no perfusion-related toxicity
  Other Names: Tecentriq; RO5541267; MPDL3280A

SUMMARY:
This is a national, single arm, phase II trial in patients with diagnosis of unresectable or advanced malignant pleural mesothelioma who experienced progression after platinum-based chemotherapy.

DETAILED DESCRIPTION:
The study includes a screening period a treatment period, a termination treatment visit ≤30 days following the last dose of the study drug, and a follow-up period. Day 1 is defined as the first day in which patients receive atezolizumab. The study is expected to enroll 36 patients.

Enrolled patients will receive a fixed dose of atezolizumab 1200 mg administered intravenously the first day of each cycle. A treatment cycle will last 21 days (± 3 days). Treatment with atezolizumab will continue until investigator-assessed loss of clinical benefit, unacceptable toxicity, investigator or participant's decision to withdraw from therapy, or death (whichever occurs first).

Treatment with atezolizumab may continue while patients experience clinical benefit based on the investigator's assessment (absence of unacceptable toxicity or symptomatic deterioration attributable to disease progression, at the discretion of the investigator after evaluating radiographic data, biopsy results [if available], and clinical status), or until unacceptable toxicity or death.

During treatment, patients treated with atezolizumab, who demonstrate evidence of clinical benefit may continue treatment with atezolizumab after meeting disease progression criteria, based on the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. The following need to be met, as specified by the protocol.

All patients must undergo tumor assessments at baseline and every 9 weeks (± 7 days) following cycle 1, day 1, regardless of treatment delays, until radiographic disease progression, as per RECIST v1.1 modified for mesothelioma, or loss of clinical benefit in patients treated with atezolizumab, who continue treatment beyond disease progression, as per RECIST v1.1, withdrawal of consent, death or study termination by principal investigator, whichever occurs first.

The study will end if all enrolled patients die, withdraw their consent, become lost to follow-up, or have been monitored during 12 months from the enrollment of the last patient, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Patients have ≥18 years of age.
* Diagnosis of malignant pleural mesothelioma histologically confirmed by certified pathologist.
* Unresectable and/or advanced disease, based on the Seventh Edition American Joint Committee on Cancer (AJCC) Cancer Staging Manual. Patients with MPM diagnosed with early disease and whose comorbidities make them ineligible for surgical procedures or who do not accept surgery treatment.
* Patients should have received at least one platinum-based treatment and should have reported progression after at least two treatment cycles.
* Disease measurable as per the Response Evaluation Criteria in Solid Tumors (RECIST) modified for mesothelioma.
* ECOG performance status ≤2.
* >12-week life expectancy.
* Patients with adequate organ function
* Patients should have recovered to grade ≤1 in all adverse events associated with previous antineoplastic therapies, excluding alopecia.
* Patients should be able to comply with protocol procedures, at the discretion of the investigator
* Patients of both genders who are potentially fertile should use effective contraceptive methods (barrier methods plus other contraceptive methods) before study entry and during their participation in the study.

Exclusion Criteria:

* Patients diagnosed with another tumor, except for treated cervical carcinoma in situ, epidermoid carcinoma, or superficial bladder cancer (Ta and Tis), or other malignancy for which healing therapy was administered within 5 years before study enrollment.
* Simultaneous participation in another study on a study drug, or if the patient participated in a study within 28 days before study treatment initiation.
* Medical history of interstitial lung disease (ILD), drug-induced interstitial disease, radiation pneumonitis that required treatment with steroids, or any sign of clinically active interstitial lung disease.
* Use of systemic immunosuppressive therapy (use of steroids with a dose >10 mg of prednisone or other immunosuppressive therapy).
* Presence of active autoimmune disease.
* Suspicion or certainty of symptomatic brain metastasis or spinal cord compression. Patients with asymptomatic and stable brain metastasis are eligible for the study.
* Pregnant or breastfeeding women. Women of childbearing potential must have a negative pregnancy test carried out within 7 days prior to treatment initiation.
* Patient previously treated with immunotherapy (PD-1/PD-L1 inhibitors).
* Major surgery within 4 weeks prior to study treatment initiation or expected major surgery during the course of the study for non-diagnostic purposes.
* Known seropositivity for human immunodeficiency virus (HIV). tory or symptoms of HIV may enter the study only if there is negative serology.
* Active tuberculosis.
* Administration of a live attenuated vaccine within 4 weeks prior to study treatment initiation or at any moment during the course of the study.
* Last chemotherapy cycle within 30 days prior to first treatment administration.
* Any unstable disease or condition that may threaten the patient's safety and/or the patient's study compliance.
* Drug addiction or clinical, psychological, or social disorders that may undermine the informed consent validity or affect compliance with protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | From the time of initial response until documented tumor progression or death, whichever occurs first (up to approximately 4 years)
  The number of subjects whose best confirmed objective response is a CR or PR, divided by the number of treated subjects

SECONDARY OUTCOMES:
Progression-free survival | Baseline up to disease progression or death, whichever occurs first (up to approximately 4 years)
  The time from the date of the start of treatment to the date of the first documented tumor progression as determined by RECIST v 1.1, or death, whichever occurs first
Duration of response | Baseline up to disease progression or death, whichever occurs first (up to approximately 4 years)
  The time from documentation of tumor response to disease progression as determined by RECIST v1.1
Overall survival | Baseline up to 1 year after treatment discontinuation
  The time from the date of the start of treatment until death from any cause
Safety of atezolizumab | Baseline up to 60 days after the last dose of the study drug or until another oncologic treatment is initiated, whichever occurs first
  The incidence of treatment-related adverse events assessed by CTCAE v4.03
Health Related Quality of Life (HRQoL) Scores | Baseline until 1 year after treatment discontinuation or death, whichever occurs first
  Change from Baseline in Health Related Quality of Life (HRQoL) Scores as Measured by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - C30 (EORTC QLQ-C30)
Patient Functioning and Symptoms Score | Baseline until 1 year after treatment discontinuation or death, whichever occurs first
  Change from Baseline in Patient Functioning and Symptoms Score as Measured by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer Module LC-13 (QLQ-LC13)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Arturo Alatorre Alexander, MD, Principal Investigator — Health Pharma Professional Research
Locations (1):
- Health Pharma Professional Research, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No